CLINICAL TRIAL: NCT06459453
Title: Effects of Kaltenborn Versus Mulligan Techniques on Pain, Range of Motion and Functional Disability in Patients With Rheumatoid Arthritis Of The Wrist.
Brief Title: Effects of Kaltenborn Versus Mulligan Techniques in Rheumatoid Arthritis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/01109
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Rheumatoid Arthritis
Keywords: : Rheumatoid arthritis, Wrist joint , Kaltenborn, Mulligan
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of the treatment arms at the begining of the trial and continue in that arm throughout the length of the trial.
Who Masked: Outcomes Assessor
Masking Description: Blinding refers to a practice where study participants are prevented from knowing certain information that may somehow influence them thereby tainting the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kaltenborn Technique (Active Comparator): Per participant was randomized to receive weekly low grade Kaltenborn manual mobilization(grade I).Any tightening of the connective tissues surrounding the joint gave (grade II) and oscillations followed by additional stretching gave (grade III).For wrist joints, Kaltenborn mobilization was performed to improve wrist flexion, extension ,radial and ulnar deviation.The duration of intervention will be 4 weeks,3 sessions per week, a total of 12 sessions will be given to the study participants.Each session will be last for 30 minutes .Conventional physical therapy will be given to the participants along with the kaltenborn mobilization.
  Interventions: Other: Kaltenborn
- Mulligan Technique (Experimental): Per participant gave concurrent application of sustained accessory mobilization applied by a therapist and an active physiological movement to end range applied by the patient . Mulligan mobilization was performed for wrist flexion and extension,(in the form of a fist)MCP joint flexion and extension,Thumb IC joint flexion and extension ,abduction and adduction of fingers.. The duration of intervention will be 4 weeks,3 sessions per week, a total of 12 sessions will be given to the study participants . Each session will last for 30 minutes .Conventional physical therapy will be given to the participants along with mulligan mobilization.
  Interventions: Other: Mulligan

INTERVENTIONS:
Other: Kaltenborn — Per participant was randomized to receive low grade Kaltenborn manual mobilization(grade I).Any tightening of the connective tissues surrounding the joint (grade II) or oscillations followed by additional stretching (grade III).Kaltenborm mobilization is performed for wrist flexion,extension,radial and ulnar deviation.The duration of intervention will be 4 weeks,3 sessions per week, a total of 12 sessions will be given to the study participants. Each session will be last for 30 minutes .Conventional physical therapy will be given to the participants along with kaltenborn.
  Arms: Kaltenborn Technique
Other: Mulligan — Per participant gave concurrent application of sustained accessory mobilization applied by a therapist and an active physiological movement to end range applied by the patient. Mulligan mobilization is performed for wrist flexion and extension(in the form of fist)MCP joint flexion and extension,Thumb IC joint flexion and extension, abduction and adduction of fingers, The duration of intervention will be 4weeks,3 sessions per week ,a total of 12 sessions will be given to the study participants .Each session will last for 30 minutes. Conventional physical therapy will be given to the participants along with conventional physiotherapy.
  Arms: Mulligan Technique

SUMMARY:
This project was a randomized control trial conducted to check the effects of kaltenborn versus mulligan techniques on pain ,range of motion and functional disability in patients with rheumatoid arthritis of the wrist The inflammatory polyarthritis that primarily affects the tiny joints is a hallmark of rheumatoid arthritis, a chronic autoimmune illness. It is characterized by synovial joint degeneration, joint swelling, and joint discomfort, which can result in disability and early death .All patients of chronic stage,convenience sampling technique was used,subjects following eligibility criteria from Shaikh zayed hospital lahore ,were randomly allocated into two groups ,baseline assessment was done.Group A participants were given Kaltenborn mobilization along with conventional physiotherapy.Group B participants were given Mulligan mobilization along with conventional physiotherapy.Post intervention assessment was done via,VAS(visual analogue scale),goniometric measurements of wrist ranges,and QUICK DASH score.3 sessions per week were given,Data was analyzed by using SPSS.

DETAILED DESCRIPTION:
Rheumatoid arthritis is among the most commonly reported problems to physicians, orthopedics and physical therapist.Even before reporting to clinics there is a long history of using over the counter pain killers.Pain avoidance behaviors let the joint stiff so much that a clinician help is sought.Most times the cause of rheumatoid arthritis is not known therefore it is term as "autoimmune disorder".There is a vast literature regarding the management of rheumatoid arthritis and yet after the decades of research there are gaps in the treatment plan.In modern age of health care it is common goal of every health care to make patient self sufficient as early as possible .The self care model has new treatment protocols All patients of chronic stage,convenience sampling technique was used, subjects following eligibility criteria from Shaikh zayed hospital lahore ,were randomly allocated into two groups ,baseline assessment was done. Group A participants were given Kaltenborn mobilization along with conventional physiotherapy .Group B participants were given Mulligan mobilization along with conventional physiotherapy. Post intervention assessment was done via,VAS(visual analogue scale),goniometric measurements of wrist ranges ,and QUICK DASH score.3 sessions per week were given,Data was analyzed by using SPSS. .This study has compared the effectiveness of kaltenborn versus mulligan mobilization on pain,range of motion and functional disabilty in patients with rheumatoid arthitis of the wrist.The current study was narrative in a way that in literature there is no comparison of two different mobilizations about treating rheumatoid arthritis.These two mobilizations were employed to see which is more effective to improve pain,range of motion and functional disability in rheumatoid arthritis of the wrist.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18 to 65 years. Patients with less than 15degrees of flexion and 30 degrees of extension.
* Male and female both are included.
* Patients with chronic RA.
* Consider only those patients with Ra factor positive. Patients with less than 10degrees of radial deviation and 15 degrees of ulnar deviation.
* Patients willing to participate in the whole treatment session and follow up.

Exclusion Criteria:

* Patients who had any mental illness (Alzheimer's, Parkinson's disease, Dementia etc)
* Patients who had any neurological deficit(paresthesia ,sensory loss, radiculopathy ,myleopathy)
* Peripheral vascular diseases.
* Any history of surgery related to upper limb.
* Patients having metal implants in the upper limbs. Patients with any other serious pathology .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-07-05 (Estimated); Study Completion 2024-08-06 (Estimated)

PRIMARY OUTCOMES:
VAS(visual analogue scale) | 4 weeks
  The visual analogue scale measures pain intensity .it consists of a 10cm line, with two end points representing 0 ('no pain')and 10('worst pain').The patient rate their current level of pain by placing a mark on the line. .
GONIOMETER | 4 weeks
  Goniometer is an instrument used to determine range of motion in patients joint .During rehabilitation, a goniometer would also be used to measure what progress has been achieved in returning back to normal range of motion.In rheumatoid arthritis of the wrist , goniometer measures the range of flexion ,extension ,radial and ulnar deviation of the wrist joint .
QUICK DASH | 4weeks
  It is the 11 item questionnaire that measures upper extremity specific symptoms and disability. It can be used to access any region of the upper extremity. The first 6 items measure the degree of difficulty in performing various physical activities and the other five items related to quality of sleeping, social activities ,daily activities and the intensity of pain and numbness.

CONTACTS AND LOCATIONS:
Overall Officials: Hajra Anwer, Principal Investigator — Riphah International University
Locations (1):
- Shaikh zayed hospital, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Maini RN, Breedveld FC, Kalden JR, Smolen JS, Furst D, Weisman MH, St Clair EW, Keenan GF, van der Heijde D, Marsters PA, Lipsky PE; Anti-Tumor Necrosis Factor Trial in Rheumatoid Arthritis with Concomitant Therapy Study Group. Sustained improvement over two years in physical function, structural damage, and signs and symptoms among patients with rheumatoid arthritis treated with infliximab and methotrexate. Arthritis Rheum. 2004 Apr;50(4):1051-65. doi: 10.1002/art.20159. PMID 15077287
- [Background] Gavrila BI, Ciofu C, Stoica V. Biomarkers in Rheumatoid Arthritis, what is new? J Med Life. 2016 Apr-Jun;9(2):144-8. PMID 27453744
- [Background] Targonska-Stepniak B, Grzechnik K, Kolarz K, Gagol D, Majdan M. Systemic Inflammatory Parameters in Patients with Elderly-Onset Rheumatoid Arthritis (EORA) and Young-Onset Rheumatoid Arthritis (YORA)-An Observational Study. J Clin Med. 2021 Mar 14;10(6):1204. doi: 10.3390/jcm10061204. PMID 33799362
- [Background] Carmona L, Villaverde V, Hernandez-Garcia C, Ballina J, Gabriel R, Laffon A; EPISER Study Group. The prevalence of rheumatoid arthritis in the general population of Spain. Rheumatology (Oxford). 2002 Jan;41(1):88-95. doi: 10.1093/rheumatology/41.1.88. PMID 11792885
- [Background] Guan CM, Beg S. Diet as a Risk Factor for Rheumatoid Arthritis. Cureus. 2023 May 20;15(5):e39273. doi: 10.7759/cureus.39273. eCollection 2023 May. PMID 37378145
- [Background] Ilan DI, Rettig ME. Rheumatoid arthritis of the wrist. Bull Hosp Jt Dis. 2003;61(3-4):179-85. PMID 15156823
- [Background] Lee KA, Min SH, Kim TH, Lee SH, Kim HR. Magnetic resonance imaging-assessed synovial and bone changes in hand and wrist joints of rheumatoid arthritis patients. Korean J Intern Med. 2019 May;34(3):651-659. doi: 10.3904/kjim.2016.271. Epub 2017 Nov 24. PMID 29166759
- [Background] Zelnio E, Taljanovic M, Manczak M, Sudol-Szopinska I. Hand and Wrist Involvement in Seropositive Rheumatoid Arthritis, Seronegative Rheumatoid Arthritis, and Psoriatic Arthritis-The Value of Classic Radiography. J Clin Med. 2023 Mar 30;12(7):2622. doi: 10.3390/jcm12072622. PMID 37048705
- [Background] Papp SR, Athwal GS, Pichora DR. The rheumatoid wrist. J Am Acad Orthop Surg. 2006 Feb;14(2):65-77. doi: 10.5435/00124635-200602000-00002. PMID 16467182
- [Background] Kurko J, Besenyei T, Laki J, Glant TT, Mikecz K, Szekanecz Z. Genetics of rheumatoid arthritis - a comprehensive review. Clin Rev Allergy Immunol. 2013 Oct;45(2):170-9. doi: 10.1007/s12016-012-8346-7. PMID 23288628
- [Background] McInnes IB, O'Dell JR. State-of-the-art: rheumatoid arthritis. Ann Rheum Dis. 2010 Nov;69(11):1898-906. doi: 10.1136/ard.2010.134684. PMID 20959326
- [Background] Korczowska I. Rheumatoid arthritis susceptibility genes: An overview. World J Orthop. 2014 Sep 18;5(4):544-9. doi: 10.5312/wjo.v5.i4.544. eCollection 2014 Sep 18. PMID 25232530
- [Background] Winchester R. The molecular basis of susceptibility to rheumatoid arthritis. Adv Immunol. 1994;56:389-466. doi: 10.1016/s0065-2776(08)60456-3. No abstract available. PMID 7521116
- [Background] Halverson PB. Extraarticular manifestations of rheumatoid arthritis. Orthop Nurs. 1995 Jul-Aug;14(4):47-50. doi: 10.1097/00006416-199507000-00009. PMID 7659452
- [Background] Markusse IM, Dirven L, Gerards AH, van Groenendael JH, Ronday HK, Kerstens PJ, Lems WF, Huizinga TW, Allaart CF. Disease flares in rheumatoid arthritis are associated with joint damage progression and disability: 10-year results from the BeSt study. Arthritis Res Ther. 2015 Aug 31;17(1):232. doi: 10.1186/s13075-015-0730-2. PMID 26321751
- [Background] Zhang C. Flare-up of cytokines in rheumatoid arthritis and their role in triggering depression: Shared common function and their possible applications in treatment (Review). Biomed Rep. 2021 Jan;14(1):16. doi: 10.3892/br.2020.1392. Epub 2020 Nov 19. PMID 33269077
- [Background] Molnar-Kimber KL, Kimber CT. Each type of cause that initiates rheumatoid arthritis or RA flares differentially affects the response to therapy. Med Hypotheses. 2012 Jan;78(1):123-9. doi: 10.1016/j.mehy.2011.10.006. Epub 2011 Nov 1. PMID 22051110
- [Background] Tanski W, Wojciga J, Jankowska-Polanska B. Association between Malnutrition and Quality of Life in Elderly Patients with Rheumatoid Arthritis. Nutrients. 2021 Apr 12;13(4):1259. doi: 10.3390/nu13041259. PMID 33921207
- [Background] Arnett FC, Edworthy SM, Bloch DA, McShane DJ, Fries JF, Cooper NS, Healey LA, Kaplan SR, Liang MH, Luthra HS, et al. The American Rheumatism Association 1987 revised criteria for the classification of rheumatoid arthritis. Arthritis Rheum. 1988 Mar;31(3):315-24. doi: 10.1002/art.1780310302. PMID 3358796
- [Background] Rydholm M, Sharma A, Jacobsson L, Turesson C. The relation between synovitis of individual finger joints and grip force over the first 5 years in early rheumatoid arthritis - a cohort study. Arthritis Res Ther. 2023 Nov 30;25(1):231. doi: 10.1186/s13075-023-03212-6. PMID 38037132
- [Background] Ajeganova S, Huizinga T. Sustained remission in rheumatoid arthritis: latest evidence and clinical considerations. Ther Adv Musculoskelet Dis. 2017 Oct;9(10):249-262. doi: 10.1177/1759720X17720366. Epub 2017 Aug 2. PMID 28974987
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of rheumatoid arthritis. Ann Rheum Dis. 1957 Dec;16(4):485-93. doi: 10.1136/ard.16.4.485. No abstract available. PMID 13498603